CLINICAL TRIAL: NCT00294957
Title: Psychological and Physiological Status of Former Prisoners of War
Status: Withdrawn | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Other Study IDs: SHEBA-05-3910-JZ-CTIL
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Assessing the psychological and physiological status of Israeli former prisoners of war (POW).

ELIGIBILITY:
Inclusion Criteria:

* Former POW

Exclusion Criteria:

* Was not defined

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Study Director — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel